CLINICAL TRIAL: NCT02221505
Title: A Phase I, Multicenter, Open-label Dose Escalation and Expansion Study of LOP628, Administered Intravenously in Adult Patients With cKit-positive Tumors and Acute Myeloid Leukemia
Brief Title: Phase 1 Study of LOP628 in Adult Patients With cKit-positive Solid Tumors and Acute Myeloid Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLOP628X2101
Record Dates: First submitted 2014-08-08; First posted 2014-08-20 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-04

CONDITIONS: cKIT-positive Solid Tumors; AML
Keywords: LOP628,; cKit,; ADC,; Antibody drug conjugates,; maytansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LOP628 - Solid Tumor (Experimental): with LOP628
  Interventions: Drug: LOP628
- LOP628 - AML (Experimental): With LOP628
  Interventions: Drug: LOP628
- LOP628 - Solid Tumor Expansion (Experimental): With LOP628
  Interventions: Drug: LOP628

INTERVENTIONS:
Drug: LOP628

SUMMARY:
LOP628 is an antibody-drug conjugate (ADC) consisting of an anti-cKit humanized IgG1/κ antibody conjugated to a maytansine payload via a non-cleavable linker.

LOP628 provides an opportunity to target cKit overexpressing tumors.

ELIGIBILITY:
Inclusion Criteria:

For patients with solid tumors:

* documented cKit-positive neoplasms
* Patient must have progressive disease as defined by any of the following:
* SCLC: patient has progressed after at least 1 prior therapy
* GIST : patient has relapsed or has refractory disease, and no further approved effective therapeutic option exists
* Patients with other cKit-positive solid tumors: patient has progressed after at least one prior line of therapy and no further approved effective therapeutic option exists
* Patient has measurable disease as per RECIST v1.1 criteria

For patients with AML:

* documented cKit-positive acute myelogenous leukemia
* Consent to newly obtained bone marrow aspirate
* Patient must have progressive disease defined as relapsed or refractory non-PML AML following standard therapy or for whom no effective therapy exists.
* Blast count < 50,000/mm3

Exclusion Criteria:

For patients with solid tumors:

* Patient has central nervous system (CNS) metastatic involvement unless the CNS metastases have been previously treated and the patient is clinically stable and on a stable dose of corticosteroids for at least 4 weeks prior to enrollment.
* Patient has the presence of other clinically significant hematologic, cardiac, respiratory, gastrointestinal, renal, hepatic or neurological conditions.
* Patient has a history of serious allergic reactions, which in the opinion of the investigator may pose an increased risk of serious infusion reactions
* Patient has been previously treated with cKit directed antibodies
* Pregnant or nursing women

For patients with AML:

* Patient has received prior allogeneic bone marrow transplant (BMT).
* Patient has the presence of other clinically significant cardiac, respiratory, gastrointestinal, renal, hepatic or neurological disease
* Patient has a history of serious allergic reactions, which in the opinion of the investigator may pose an increased risk of serious infusion reactions
* Patient has been previously treated with cKit directed antibodies
* Pregnant or nursing women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-12; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Incident rate of dose limiting toxicities (DLTs) | Month 12
  To estimate the maximum tolerated dose/recommended dose for expansion (MTD/RDE)

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAE) | 30 months
  Characterize the safety and tolerability of LOP628
Severity of adverse events (AEs) and serious adverse events (SAEs) | 30 months
  Characterize the safety and tolerability of LOP628
Serum PK parameters (AUC, Cmax, Tmax, and half-life) | 30 months
  To characterize the pharmacokinetic profile of LOP628
Serum concentration vs. time profiles | 30 months
  To characterize the pharmacokinetic profile of LOP628.
Overall response rate (ORR) | 30 months
  To assess the preliminary anti-tumor activity of LOP628
Duration of response (DOR) | 30 months
  To assess the preliminary anti-tumor activity of LOP628
Progression Free Survival (PFS) | 30 months
  To assess the preliminary anti-tumor activity of LOP628
Disease Control Rate (DCR) at 4 months | 4 months
  To assess the preliminary anti-tumor activity of LOP628
Best overall response (BOR) | 30 months
  To assess the preliminary anti-tumor activity of LOP628 in patients
Best Overall Response (AML) | 30 months
  To assess the preliminary anti-tumor activity of LOP628
Duration of response (DOR) (AML) | 30 months
  To assess the preliminary anti-tumor activity of LOP628
Event Free Survival (EFS) (AML) | 30 months
  To assess the preliminary anti-tumor activity of LOP628

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (4):
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Leuven, Belgium
- Novartis Investigative Site, Leiden, Netherlands
- Novartis Investigative Site, Barcelona, Catalonia, Spain